CLINICAL TRIAL: NCT02074384
Title: Understanding Patient and Provider Glucose Reporting Preferences in Type 1 Diabetes: Cloud Based Ambulatory Glucose Profile (AGP)
Brief Title: Patient and Provider Glucose Reporting Preferences Ambulatory Glucose Profile (AGP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 04356-14-A
Record Dates: First submitted 2014-02-25; First posted 2014-02-28 (Estimated); Results first posted 2016-01-01 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2015-10

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Glucose Self-Monitoring; Nurse Clinicians

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Continuous Glucose Monitoring (Other): Participants will wear Continuous Glucose Monitoring for two weeks.
  Interventions: Device: Continuous Glucose Monitor
- Self Monitoring Blood Glucose (Other): Participants will self test for two weeks.
  Interventions: Device: Self Monitoring Blood Glucose
- Clinicians (Other): Clinicians completing study visits.
  Interventions: Other: Clinician

INTERVENTIONS:
Device: Continuous Glucose Monitor — CGM device for measurement of interstitial glucose on a 24/7 continuous cycle.
  Other Names: Dexcom G4 professional version Continuous Glucose Monitor
  Arms: Continuous Glucose Monitoring
Device: Self Monitoring Blood Glucose — Participants will use their own SMBG device.
  Arms: Self Monitoring Blood Glucose
Other: Clinician — Survey of clinicians after study visits
  Arms: Clinicians

SUMMARY:
International Diabetes Center (IDC) proposes a preference and usability study of glucose data acquisition and reporting, evaluating streamlined standardized cloud-based glucose reporting including work flow as well as patient and clinician preference at Type 1 Diabetes (T1D) Exchange sites to enhance standard Ambulatory Glucose Profile (AGP) reporting. This phase 2 project assesses the efficacy of standardized glucose data report generation and preferred report presentation format; both are necessary to increase use of continuous glucose monitoring (CGM) data to improve care processes and outcomes for Type 1 diabetes.

DETAILED DESCRIPTION:
Patient participation in diabetes treatment has relied upon episodic self-monitoring of blood glucose (SMBG). SMBG assists patients and clinicians with adjustments of insulin, identification of hypoglycemia, nutritional intake and activity in order to optimize diabetes control. SMBG however is subject to bias dependent upon the testing frequency and timing. In contrast, continuous glucose monitoring (CGM) systems capture continuous 24-hour glucose data uninterrupted and unbiased. It provides valuable information about daily/nightly alterations in glucose patterns. Unfortunately SMBG, CGM and insulin pump devices have proprietary software with unique data standards, acquisition methods, reports, and graphic displays. These differences make evaluation and comparison of SMBG or CGM data difficult for clinicians and patients. IDC created an Ambulatory Glucose Profile (AGP) report to reduce challenges of device specific reports through a standardized report which is produced from any device with streamlined graphic displays of glucose trends.

The phase 1 project (2012), gathered expert stakeholders (clinical, research, industry, patients) who validated data standards and recommended changes to the CGM-AGP reports. These changes are now integrated into a secure cloud-based infrastructure for AGP reporting.

Phase 2 of this project is a usability and preference study of glucose reporting systems. It will include an in depth study of 6 T1D Ex clinical sites. The T1D Exchange Clinic Network was formed to support the development of a large registry of adults and children with type 1 diabetes for the purpose of conducting multiple studies proposed by T1D Exchange investigators, and other researchers, patients, and companies.

The 6 sites will be selected for an in-depth study utilizing middleware data collection services (Diasend or SweetSpot) to facilitate efficient collection of data from diverse devices. These middleware solutions integrate with the captūrAGP system to automatically produce an AGP report. These sites will test the feasibility of AGP cloud reporting while collecting patient and clinician opinions on report preference. All 6 sites participating in phase 2 will collect patient and clinician preference measures. Two study sites will undergo time in motion (TIM) measurement and workflow mapping of current process. This TIM sub-study includes workflow mapping of current and cloud-based processes utilizing Toyota Lean (Kaizen) methodology. Sites 3 - 6 will receive enhanced designs through the adaptive trial method with learnings applied from sites 1 and 2.

A key deliverable of this study is patient and clinician insight into their utilization of CGM reporting technologies. Recognizing that adoption of technology is often stymied by time constraints, report reliability and ease of interpretation, these variables will be examined. The goal of phase 2 is to analyze the viability of standard reporting and to evaluate preference (patient and clinicians) for and perceived value of different types of glucose pattern reports (AGP vs. device) including clinical practice time saved.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetics

Exclusion Criteria:

* Less than the age of 7
* Non-English Speaker

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bergenstal, MD, Principal Investigator — Park Nicollet; Deborah Mulllen, PhD, Principal Investigator — Park Nicollet
Locations (7):
- United States (7):
  - Eda Cengiz, New Haven, Connecticut
  - Larry Deeb, Tallahassee, Florida
  - Henry Ford, Detroit, Michigan
  - Park Nicollet International Diabetes Center, Minneapolis, Minnesota
  - The Diabetes Center, PLLC, Ocean Springs, Mississippi
  - St. Vincent's, Billings, Montana
  - Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinicians: Clinicians completing study AGP visits.
Period: Overall Study
Arm/Group | Continuous Glucose Monitoring | Self Monitoring Blood Glucose | Clinicians
Started | 74 | 70 | 17
Completed | 74 | 70 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Clinicians: Clinicians completing the study visits.
- Total: Total of all reporting groups
Arm/Group | Continuous Glucose Monitoring | Self Monitoring Blood Glucose | Clinicians | Total
Number analyzed (Participants) | 74 | 70 | 17 | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 32 | 0 | 72
  Between 18 and 65 years | 34 | 36 | 17 | 87
  >=65 years | 0 | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.0 (14.5) | 28.8 (18.7) | NA (NA) — Not collected | 26.4 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 38 | NA — Not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | 40 | 32 | NA — Not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 74 | 70 | 17 | 161

OUTCOME MEASURES:

1. Primary Outcome: Portion of Study Participants Reporting Greater Utility From AGP vs. Traditional Glucose Data Reports
Description: Patients will use either SMBG or CGM for a two week period following their screening visit. At the end of the two week period they will return to the study site to download their device and have an AGP report printed. They will then complete a preference and utility survey.
Time Frame: At the end of the two week SMBG or CGM period
Measure: Number; unit: participants
Arm/Group | Continuous Glucose Monitoring | Self Monitoring Blood Glucose | Clinicians
Number analyzed (Participants) | 70 | 70 | 17
participants | 35 | 29 | 10

ADVERSE EVENTS:
Time Frame: 1 year and 6 months
Arm/Group | Continuous Glucose Monitoring | Self Monitoring Blood Glucose | Clinicians
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70 | 0/17
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70 | 0/17

LIMITATIONS AND CAVEATS:
This is a survey of patient and clinician preference and as such is subject to traditional survey biases (social desirability, hawthorne effect, etc.).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No